CLINICAL TRIAL: NCT03507985
Title: Attention and Memory Disorders Related to Acute Morphine
Acronym: MEMOMORPH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0144; 2018-A00991-54 (Other: ID-RCB)
Record Dates: First submitted 2018-04-20; First posted 2018-04-25 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Memory Disorders
Keywords: morphine; attention disorders
MeSH Terms: conditions — Memory Disorders; Cognition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The exposed group: The exposed group where patients receive morphine analgesia The patient will realise two tests evaluating memory and attention, for the first at the inclusion visit after giving his consent, and in a second time during the follow up visit 15 days or 1 month later.
  Interventions: Other: Two tests evaluating memory and attention
- The unexposed group: The unexposed group where patients receive 1 +/- 2-stage analgesia is non-opioid analgesics.
  The patient will realise two tests evaluating memory and attention, for the first at the inclusion visit after giving his consent, and in a second time during the follow up visit 15 days or 1 month later.
  Interventions: Other: Two tests evaluating memory and attention

INTERVENTIONS:
Other: Two tests evaluating memory and attention — The patient will perform two tests assessing memory and attention:
  Regarding attention, the test used will be the Stroop Color Word Test, developed to measure visual selective attention, cognitive flexibility and inhibition.
  For memory, the test used will be Rey's 15 words test. It provides an indicative standard for the evaluation of episodic verbal memory and learning abilities. This test was compared to the 16-item (18) free recall / booster test in normal aging and Alzheimer's dementia, and although it was more difficult, it . Since it allowed for the classification of participants from both groups without overlap

SUMMARY:
The aim of the study is to determine if there are attention disorders related to acute morphine use in single-traumatized patients and after that the investigators will determine whether there are immediate memory problems associated with acute morphine withdrawal in single-traumatized patients.

From a biochemical point of view, the analgesic effects of morphine and the central side effects appear to be two different dimensions of the action of morphine, each related to a metabolite. Regarding acute attention, it is difficult to differentiate attention deficit disorder due to pain or due to morphine.

Two tests have been validated in the literature to evaluate attention and memory: the 15 words of Rey and the Stroop Color Word test. The investigators will use these two tests in this study.

DETAILED DESCRIPTION:
Morphine is a powerful analgesic used in chronic non-neuropathic cancerous (Walsh) and non-cancerous (Zenz et al) pain and for the relief of acute trauma pain, for example.

It is know that morphine as well as pain can cause cognitive disorders but the pain seems to slow down the reaction time whereas morphine has an action on the long-term memory (Lorenz J et al). According to an experimental study on rats, low dose morphine (equivalent to that present in the human brain) does not cause long-term memory problems, as opposed to a higher dose. In healthy volunteers, a single dose of morphine gives little cognitive and psychomotor dysfunction (Hank et al). After 12 months of taking oral morphine, no cognitive dysfunction is detected, with even some improvement for some functions related to stopping pain. More recently, it has been shown that long-term morphine use causes spatial memory disturbances and that these are probably due to extracellular adenosine accumulation.

This work suggests that acute morphine could lead to memory and attention disorders. This would therefore result in intrinsic impairment of the cognitive abilities of the patient and thus an alteration of his understanding in the explanations given concerning a possible surgical intervention, the risks and benefits of it.

The purpose of the study is to assess the patient's attention and memory skills after acute morphine use. In order to know their initial capacities, the tests are also done remotely outside the influence of the analgesic drugs given to the emergency services. The two practical tests, the Stroop Color Word Test and Rey's 15-word test, are easily performed tests in an emergency context and validated in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Mono traumatized (suspicion of bone fracture) without vital distress, neurological, cardio-circulatory or pulmonary involvement
* Analgesia obtained, defined by a pain score on a numerical scale ≤ 3/10 at the end of the treatment
* Patient to be re-convened for plaster repair, control radiography or specialized consultation in the month following inclusion.
* Patients presenting in an emergency department of Toulouse University Hospital

Exclusion Criteria:

* Patients with vital distress, whatever the cause,
* Traumatized cranial,
* pre-existing labeled attention disorders (eg, diagnosed hyperactivity),
* Pre-existing memory disorders labeled (eg, dementia)
* Use of opioid analgesics other than morphine in the care of these patients
* Chronic opiate users (licit or illicit)
* Psychiatric disorders
* Acute alcohol poisoning, voluntary drug poisoning or not, acute intoxication by drugs
* Visual disorders (colorblind ..), patients who can not read

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two groups of patients :
  The exposed group where patients receive morphine analgesia The unexposed group where patients receive stage 1 +/- 2 analgesia is non-opioid analgesics.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The comparison of acute attention deficit according to the exposed or unexposed patient. | 1 month
  The primary endpoint selected is the comparison of acute attention deficit according to the exposed or unexposed patient.
  For each patient, the investigators will calculate the percentage of deficit between the Stroop Color Word test result at inclusion and at follow-up divided by the tracking score. This acute deficit is expressed as a percentage.
  The primary endpoint selected is the comparison of acute attention deficit according to the exposed or unexposed patient.

SECONDARY OUTCOMES:
The comparison of the acute memory deficit according to the exposed or unexposed nature of the patient | 1 month
  The secondary endpoint chosen is the comparison of the acute memory deficit according to the exposed or unexposed nature of the patient.
  For each patient, the aim is to calculate the percentage of deficit between the test result of the 15 words of Reys test at inclusion and during the follow-up divided by the tracking score. This acute deficit is expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Bounes, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No